CLINICAL TRIAL: NCT06064162
Title: A Pilot Study of Intravenous, Subanesthetic Dose of Ketamine Versus Placebo, A Crossover Design, for Multiple Sclerosis Related Fatigue
Brief Title: Ketamine for MS Fatigue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alta Bates Summit Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REDI2022MS
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: MS related Fatigue
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (active treatment) (Active Comparator): dose of 0.5 mg/kg intravenously over 40 minutes on day 1
  Interventions: Drug: ketamine
- Saline (placebo treatment) (Placebo Comparator): Placebo (saline solution) over 40 minutes on day 1
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — 60mg (.5mg/kg over 40 minutes intravenously)
  Other Names: Ketalar

SUMMARY:
The purpose of this study is to see whether using ketamine to increase glutamate in the prefrontal cortex can reduce Multiple Sclerosis (MS) related fatigue. The investigator proposes a prospective, crossover, randomized, placebo-controlled study to assess the efficacy and safety of low, single dose Ketamine, to assess its efficacy and safety in patients with MS-related fatigue.

DETAILED DESCRIPTION:
The study treatment is designed in two 28-day cycles: for each cycle, participants will receive study infusion on Day 1 and complete follow-up visits during Days 7 and 28. Participants are randomized 1:1 to receive either ketamine (active treatment) or saline solution (placebo treatment) for their first infusion. They will not be blinded to their study assignment: the study doctor will disclose their assigned treatment group.

After their first infusion cycle, participents will crossover to the other treatment group. Worded differently, if a participant received ketamine during their first infusion, they will receive placebo treatment during their second infusion. Conversely, if a participant received saline treatment during their first infusion, they will receive ketamine during their second infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Female and Male patients with any form of CDMS ages 18-65 inclusive
2. Report fatigue which is interfering with QOL
3. Able and willing to sign informed consent
4. Stable on DMT for at least 3 months prior to baseline visit
5. Not experiencing an MS relapse within 90 days prior to baseline visit.
6. Must agree to practice an acceptable method of contraception
7. Experiencing significant fatigue due to MS (MFIS of ≥10)

Exclusion Criteria:

1. Allergy to Ketamine
2. Taking medications which may interact with ketamine
3. Change in DMT within 3 months prior to baseline visit
4. MS relapse within 90 days of the baseline visit
5. Confirmed diagnosis of untreated Sleep Apnea
6. Confirmed diagnosis of periodic limb movement disorder
7. Serious infection in the 30 days prior to baseline visit.
8. Patients with significant comorbid conditions:

   1. Untreated hypertension (SBP>160, DBP>100 at baseline)
   2. Liver disease
   3. Significant renal disease
   4. History of cardiac arrhythmia
   5. Any comorbidities which at the opinion of the investigators post undue risk
9. Current alcohol or drug abuse
10. Participation in another interventional clinical trial in the past 3 months.
11. Pregnant or lactating
12. Any condition which in the opinion of the investigators will cause safety concerns for the patient, or inability to comply with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Improve Fatigue Scores | 28 days post study drug infusion
  a statistically significant change in the level of fatigue score as measured by the Multiple Schlerosis fatigue scales: Modified Fatigue Impact Scale (MFIS) between baseline and day 28 post study drug infusion. Rating scale is 0 to 4 with 0 being "never" and 4 being "almost always."

SECONDARY OUTCOMES:
Improve Quality of Life | Between baseline and day 28
  A statistically significant change in the patient's quality of life as measured by Functional Index for Living with Multiple Sclerosis (FILMS) between baseline and day 28. Score is rated 1 to 5 with 1 being "bad" and 5 being "good."

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Soneji, MD, Principal Investigator — Sutter East Bay Medical Foundation
Locations (1):
- Alta Bates Summit Medical Center, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzgerald KC, Morris B, Soroosh A, Balshi A, Maher D, Kaplin A, Nourbakhsh B. Pilot randomized active-placebo-controlled trial of low-dose ketamine for the treatment of multiple sclerosis-related fatigue. Mult Scler. 2021 May;27(6):942-953. doi: 10.1177/1352458520936226. Epub 2020 Jul 7. PMID 32633662
- [Background] Saligan LN, Farmer C, Ballard ED, Kadriu B, Zarate CA Jr. Disentangling the association of depression on the anti-fatigue effects of ketamine. J Affect Disord. 2019 Feb 1;244:42-45. doi: 10.1016/j.jad.2018.10.089. Epub 2018 Oct 6. PMID 30312839
- [Background] Induruwa I, Constantinescu CS, Gran B. Fatigue in multiple sclerosis - a brief review. J Neurol Sci. 2012 Dec 15;323(1-2):9-15. doi: 10.1016/j.jns.2012.08.007. Epub 2012 Aug 27. PMID 22935407
- [Background] Kos D, Kerckhofs E, Nagels G, D'hooghe MB, Ilsbroukx S. Origin of fatigue in multiple sclerosis: review of the literature. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):91-100. doi: 10.1177/1545968306298934. Epub 2007 Apr 4. PMID 17409388
- [Background] Stankoff B, Waubant E, Confavreux C, Edan G, Debouverie M, Rumbach L, Moreau T, Pelletier J, Lubetzki C, Clanet M; French Modafinil Study Group. Modafinil for fatigue in MS: a randomized placebo-controlled double-blind study. Neurology. 2005 Apr 12;64(7):1139-43. doi: 10.1212/01.WNL.0000158272.27070.6A. PMID 15824337
- [Background] Asano M, Finlayson ML. Meta-analysis of three different types of fatigue management interventions for people with multiple sclerosis: exercise, education, and medication. Mult Scler Int. 2014;2014:798285. doi: 10.1155/2014/798285. Epub 2014 May 14. PMID 24963407
- [Background] Nourbakhsh B, Revirajan N, Morris B, Cordano C, Creasman J, Manguinao M, Krysko K, Rutatangwa A, Auvray C, Aljarallah S, Jin C, Mowry E, McCulloch C, Waubant E. Safety and efficacy of amantadine, modafinil, and methylphenidate for fatigue in multiple sclerosis: a randomised, placebo-controlled, crossover, double-blind trial. Lancet Neurol. 2021 Jan;20(1):38-48. doi: 10.1016/S1474-4422(20)30354-9. Epub 2020 Nov 23. PMID 33242419
- [Background] Broicher SD, Filli L, Geisseler O, Germann N, Zorner B, Brugger P, Linnebank M. Positive effects of fampridine on cognition, fatigue and depression in patients with multiple sclerosis over 2 years. J Neurol. 2018 May;265(5):1016-1025. doi: 10.1007/s00415-018-8796-9. Epub 2018 Feb 20. PMID 29464379
- [Background] Meca-Lallana V, Branas-Pampillon M, Higueras Y, Candeliere-Merlicco A, Aladro-Benito Y, Rodriguez-De la Fuente O, Salas-Alonso E, Maurino J, Ballesteros J. Assessing fatigue in multiple sclerosis: Psychometric properties of the five-item Modified Fatigue Impact Scale (MFIS-5). Mult Scler J Exp Transl Clin. 2019 Nov 9;5(4):2055217319887987. doi: 10.1177/2055217319887987. eCollection 2019 Oct-Dec. PMID 31741743
- [Background] Wesson JM, Cooper JA, Jehle LS, Lockhart SN, Draney K, Barber J. The functional index for living with multiple sclerosis: development and validation of a new quality of life questionnaire. Mult Scler. 2009 Oct;15(10):1239-49. doi: 10.1177/1352458509107019. Epub 2009 Sep 8. PMID 19737850
- [Background] Beard C, Hsu KJ, Rifkin LS, Busch AB, Bjorgvinsson T. Validation of the PHQ-9 in a psychiatric sample. J Affect Disord. 2016 Mar 15;193:267-73. doi: 10.1016/j.jad.2015.12.075. Epub 2015 Dec 31. PMID 26774513
- See also: National Multiple Sclerosis Society — https://www.nationalmssociety.org/